CLINICAL TRIAL: NCT04312724
Title: MSS - Clinical Investigation An Investigation of a New Manufacture Technique of a Trans-femoral Socket and Its Function for Amputees.
Brief Title: An Investigation Into a New Manufacture Technique of Trans-femoral Sockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP2017122866
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Amputation
Keywords: Trans-femoral stump mobility pain usability service socket

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Clinical need (Active Comparator): Participants enrolled that require a new socket.
  Interventions: Device: Direct Socket TF
- No clincal need (Experimental): Participants enrolled that do not require a new socket
  Interventions: Device: Direct Socket TF

INTERVENTIONS:
Device: Direct Socket TF — The device is Class I, a low-risk product, and is a further development of a well-established technology. Össur Direct Socket (DS) technology has been on the market since 1996 (ICEX first generation) for the manufacture of leg prosthesis. This prosthetic socket for trans-femoral amputees (referred hereby to as DS-TF) has the same basic functional design as the Direct Socket (MSS) for trans-tibial amputees (referred hereby to as DS-TT) that is available on the market today in addition to the newly added silicon brim.
  A prosthetic socket is a non-invasive, non-sterile, single user reusable device, which is used as part of prosthetic system. The aspect of the prosthesis that is in direct physical contact with the amputee is usually not the socket, to which a prosthesis is connected to, but the liner that serves as an interface between the amputee and the rest of the prosthesis. An amputee typically wears a prosthesis and thereby utilizes a socket, for up to 18 hours a day.
  Other Names: DS-TF; DS Trans-femoral

SUMMARY:
The investigation will be of a single group prospective pre/post design with follow up at 6 weeks (6WFU) and 6 months (6MFU); comparing to outcomes at baseline (BL).

Device(s) being tested: Interchangeably: Direct Socket TF; DS-TF; DS Trans-femoral.

The DS-TF is a trans-femoral (TF) set-up of the currently marketed trans-tibial version. It is not marketed in the USA and has not been registered with the FDA.

The comparator is the current socket the subject is using when enrolled in the study.

Subjects recruited: Minimum 50

Inclusion criteria:

50Kg< body weight < 160Kg Cognitive ability to understand all instructions and questionnaires in the study; Patients who have undergone a transfemoral amputation > 1 year post amputation Older than 18 years Willing and able to participate in the study and follow the protocol Circular dimension of 40-65 cm at the crotch Residual limb length at least 20 cm from ischium to distal end Currently using a prosthetic liner Locking users that can successfully be fitted with Iceross® Transfemoral Locking, OR Seal-In users that can successfully be fitted with either Iceross Seal-In® X5 TF or Iceross Transfemoral Seal-In®

Exclusion criteria: 50Kg> body weight > 160Kg Users with cognitive impairment Patients who have undergone a transfemoral amputation <1 year post amputation Younger than 18 years Not a prosthetic ambulator, uses only the prosthesis for cosmetic reasons Circular dimension of less than 40 cm or greater than 65 cm at the crotch Residual limb length less than 20 cm from ischium to distal end Currently not using a prosthetic liner

DETAILED DESCRIPTION:
The test will be a single group prospective pre/post design. Amputees are a small proportion of the general population. The population group specified in the inclusion/exclusion criteria is a further subsample of amputees. For practical reasons, i.e. to achieve statistical power, it is therefore more feasible to use within-subject comparison rather than creating study arms to compare. Furthermore, as mobile amputees generally have and use a prosthetic device for their daily activities, within-comparison is feasible comparing to the subjects' previous device.

All investigational activities will be conducted at prosthetic out-patient clinics.

As stated above the primary endpoint is successful use rate, see Table 2, and the secondary endpoints are listed in the table from B-H in that respective order of significance. See previous chapter on objectives and hypothesis and Table 2 for rationale.

Drop-outs and withdrawals will not be replaced.

Equipment required for each subject:

* Pen/pencil
* Printed out instruments
* Investigational device: Materials for making DS-TF socket o Designated locking or seal-in liner to be fitted with the socket

Additionally, each LPI or LCI will have access to:

* Equipment for DS-TF socket manufacturing
* iPad with the Össur ProApp installed for data collection The equipment used does not require specific monitoring, maintenance or calibration procedures.

The purpose of the study is to evaluate in a cohort the time it takes to manufacture and delivery (lead time) of a definitive prosthesis (definition of finished prosthetic leg is, a prosthesis that is individually tailored and able to be used both indoors and outdoors, with the maximum weight on the patient equivalent to 160 kg). The existing prosthesis is to be evaluated as well as the new socket. The evaluation of function will take place at baseline, 6 weeks and 6 months after deliverance.

The following outcome instruments will be used:

• At all three study evaluation points; initial fitting, 6 wees and 6 months:

* OPUS (LEFS, CSD, CSS) https://www.sralab.org/rehabilitation-measures/orthotics-prosthetics-users-survey
* ProAMP (to test the current function with prosthesis)
* EQ-5D (for life quality)
* Socket Comfort Score (SCS)
* CLASS - socket fit
* Plus-M
* ABC
* TUG

Cost of fitting, to all parties, will be collected and reported. Whatever the outcome of the study will be, it will be very informative for healthcare systems, both payers and providers, and manufacturer of equipment for amputees.

The total time required to implement the full clinical investigation is expected to be approximately 26 months. Each individual subject is expected to participate in the clinical investigation for a minimum of 6 weeks, up to 6 months. The estimated time needed to include the required number (enrolment period) is 20 months.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive ability to understand all instructions and questionnaires in the study.
* Patients who have undergone a trans-femoral amputation > 1 year post amputation.
* Willing and able to participate in the study and follow the protocol.
* Circular dimension of 40-65 cm at the crotch.
* Residual limb length at least 20 cm from ischium to distal end.

Exclusion Criteria:

* 50Kg > body weight > 160Kg
* Users with cognitive impairment
* Not a prosthetic ambulator, uses only the prosthesis for cosmetic reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
OPUS | 6 months
  Patient Self report. Paper based. Evaluation of service and device.
CLASS | 6 months
  Amputee Self-report: socket quality evaluation (comfort, pain, stability, aesthetics); collected with ProApp.
AmpPro | 6 months
  CPO evaluation of amputee, objective scoring: activity/mobility; collected with ProApp.
PLUS-M | 6 months
  Amputee Self-report: activity/mobility; collected with ProApp.
EQ-5D | 6 months
  Amputee self report: QoL, paper based.
ABC | 6 months
  Amputee self report: Activity-Balance Confidence scale; collected with ProApp.
TUG | 6 months
  Activity: Timed up and go; collected with ProApp.
CPO usability | 6 months
  In-house generated instrument; paper based

SECONDARY OUTCOMES:
Observation log | Baseline only
  Timing and documentation on how the DS-TF is fitted.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Pratt, CPO, Principal Investigator — Össur Iceland ehf
Locations (16):
- United States (16):
  - Alabama Artificial Limb Specialists, Mobile, Alabama
  - Alabama Artificial Limb Specialists, Montgomery, Alabama
  - Alabama Artificial Limb Specialists, Opelika, Alabama
  - Van Der Watt Prosthetics & Orthotics, Greenwood, Arkansas
  - Tillges Certified Orthotic Prosthetic Inc, Maplewood, Minnesota
  - Sampson's Prosthetics Lab, Albany, New York
  - Sampson's Prosthetics Lab, Schenectady, New York
  - Eastside Orthotics and Prosthetics, Portland, Oregon
  - Union Orthotics & Prosthetics Co, Cranberry Township, Pennsylvania
  - Union Orthotics & Prosthetics Co, East Rochester, Pennsylvania
  - Union Orthotics & Prosthetics Co, Greensburg, Pennsylvania
  - Union Orthotics & Prosthetics Co, Pittsburgh, Pennsylvania
  - Victory Orthotics and Prosthetics Inc., Johnson City, Tennessee
  - Victory Orthotics and Prosthetics Inc., Kingsport, Tennessee
  - Victory Orthotics and Prosthetics Inc., Knoxville, Tennessee
  - Virginia Prosthetics and Orthotics, Roanoke, Virginia